CLINICAL TRIAL: NCT04240184
Title: Physical and Psychosocial Work Environmental Risk Factors of Low-back Pain
Acronym: IRMA21
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: IRMA21
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Musculoskeletal Disorders; Stress
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Physical workload — Cohort study - The specific study aims are to investigate 1) exposure-response associations between quantity of occupational lifting and short-term (day-to-day) changes in LBP, 2) the influence of accumulated workdays and rest days during a working week on LBP, 3) long-term association between occupational lifting exposure and LBP when assessed over 1 year, and 4) the role of psychological and social factors on the above associations.

SUMMARY:
BACKGROUND:

Musculoskeletal disorders, and in particular low-back pain (LBP), are common among blue collar workers. In the work environment, both physical- and psychosocial risk factors exist. Working in warehouses in Denmark involve large quantities of occupational lifting, high work pace and a low degree of influence at work. This study investigates both acute and long-term associations between physical- and psychosocial work environmental factors and risk of LBP in warehouse workers. The specific study aims are to investigate 1) exposure-response associations between quantity of occupational lifting and short-term (day-to-day) changes in LBP, 2) the influence of accumulated workdays and rest days during a working week on LBP, 3) long-term association between occupational lifting exposure and LBP when assessed over 1 year, and 4) the role of psychological and social factors on the above associations.

METHODS:

The present study is designed as a 1-year prospective cohort study that will examine full-time warehouse workers from up to five retail chains in Denmark. Study aims 1 and 2 will be addressed using objective data based on company records with information on weight of all the goods handled by each warehouse worker during every single workday for 3 weeks. During this period, each worker will reply to text messages received before and after every workday (also on days off work) in which study participants will score their pain in the low back, bodily fatigue and perceived mental stress (scale 0-10). Long-term pain development is assessed using questionnaire surveys before and after 1 year. Further, pressure pain threshold (PPT) will be measured for selected trunk extensor muscles in approximately 50 workers using algometry along with measurements of maximal trunk extensor strength. Associations are modelled using linear mixed models with repeated measures between variables and LBP controlled for relevant confounders.

DISCUSSION:

This study provides knowledge about the acute and long-term associations between physical- and psychosocial work environmental factors and LBP. The obtained data will have the potential to provide recommendations on improved design of the working week to minimize the risk of LBP among warehouse workers, and may potentially enable to identify a reasonable maximum lifting threshold per day (ton lifted/day).

ELIGIBILITY:
Inclusion Criteria:

* working ≥30 h per week in a registered retail industry warehouse
* ability to read and understand Danish or English,
* ≥18 years of age.

Exclusion Criteria:

* Hypertension > 160/100 mmHg

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Enrolled study participants will receive a baseline questionnaire by e-mail that will address various aspects of physical-, psychological and social work environment and health. The questionnaire will also comprise an invitation to participate in a text message survey. Participants recruited for the text message survey will receive a SMS text message before and after every workday for 3 full weeks (21 days) to rate the magnitude of pain in their low back, and to score their current level of perceived physical fatigue and mental stress. During the same 3-week study period, section leaders at the warehouses will provide company records about the workload of each participating warehouse worker (goods handled by each worker, weight of the goods) along with a working schedule for each worker. One year after responding to the baseline questionnaire, the participant will be receiving a follow-up questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Short-term LBP | 21 days
  exposure-response associations between quantity of occupational lifting and short-term (day-to-day) changes in LBP
Accumulated workdays and LBP | 21 days
  the influence of accumulated workdays and rest days during a working week on LBP
Long-term LBP | 1 year
  Long-term association between occupational lifting exposure and LBP when assessed over 1 year

SECONDARY OUTCOMES:
Psychosocial influence on LBP | 21 days
  The role of psychological and social factors on outcome 1, 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Lars L Andersen, PhD, Study Director — National Research Centre for the Working Environment, Denmark; Runi Blafoss, MSc, Principal Investigator — National Research Centre for the Working Environment, Denmark
Locations (1):
- National Research Centre for the Working Environment, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No